CLINICAL TRIAL: NCT03310671
Title: Aortic Stenosis in Subjects With Heterozygous Familial Hypercholesterolemia on Prolonged Treatment With Statins
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Principal Investigator, Fernando Civeira, Instituto Aragonés de Ciencias de la Salud, Instituto Aragones de Ciencias de la Salud
Other Study IDs: C.I.PI17/0256
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Aortic Stenosis; Arteriosclerosis; Familial Hypercholesterolemia; Conventional Transthoracic Echocardiogram
MeSH Terms: conditions — Aortic Valve Stenosis; Arteriosclerosis; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASES: Cases:
  * Age ≥ 65 years at the time of cardiac ultrasound
  * Genetically diagnosed HFH or in a first-degree relative
  * History of hypercholesterolemia with LDLc levels> 220 mg / dL without lipid-lowering treatment
  Interventions: Procedure: Echocardiogram
- Controls: * Genetically Similar
  * Siblings of the normocholesterolemic case, defined by LDLc <190 mg / dl without lipid-lowering treatment.
  * In the absence of available siblings, first cousins may be included.
  * In the presence of several siblings available, the same sex will be included,
  * Environmentally similar
  * Stable partner of the case with cohabitation> 25 years
  Interventions: Procedure: Echocardiogram

INTERVENTIONS:
Procedure: Echocardiogram — Conventional transthoracic echocardiogram by an echocardiographer trained to perform and centered on aortic valve
  Pick up from:
  * Mean transvalvular pressure gradient
  * Aortic valve
  * Aortic valve opening area
  * Aortic valve opening area adjusted for body mass index
  * Bicuspid or tricuspid aorta
  * Thickness of the upper valve> 3 mm

SUMMARY:
Aortic stenosis (AE) is a disease that has been increasing steadily in recent years in most countries, including Spain.Risk factors for the development of AE include age, hypercholesterolemia, diabetes mellitus and arterial hypertension, the classic risk factors for the development of atherosclerosis. However, lipid-lowering therapy with statins and ezetimibe has not been shown to reduce the risk of long-term progression of AE by unknown mechanisms. All this suggests that subjects with HFhe have a high risk of developing AD, which has not been shown by the high coronary mortality in this population that precedes aortic calcification

DETAILED DESCRIPTION:
The study includes a single clinical visit with collection of clinical data, blood extraction and the performance of a transthoracic echocardiogram. This visit may be made on different days, but always within 30 days of signing the informed consent.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Age ≥ 65 years at the time of cardiac ultrasound
* Genetically diagnosed HFH or in a first-degree relative
* History of hypercholesterolemia with LDLc levels> 220 mg / dL without lipid-lowering treatment

Controls:

* Genetically Similar
* Siblings of the normoccholesterolemic case, defined by LDLc <190 mg / dl without lipid-lowering treatment.
* In the absence of available siblings, first cousins may be included.
* In the presence of several siblings available, the same sex will be included,
* Environmentally similar
* Stable partner of the case with cohabitation> 25 years * Each case will have at least one control.

Exclusion Criteria:

- Personal history of cardiac rheumatic disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Genetically diagnosed HFH or in a first-degree relative
  - History of hypercholesterolemia with LDLc levels> 220 mg / dL without lipid-lowering treatment
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-07-18 (Estimated); Study Completion 2018-07-18 (Estimated)

PRIMARY OUTCOMES:
Differences in age-adjusted prevalence of EA assessed by transthoracic echocardiography between cases and controls | 1 YEAR

SECONDARY OUTCOMES:
Differences in age-adjusted prevalence of AD assessed by transthoracic echocardiography between cases and controls | 1 YEAR
Difference in aortic surface between cases and controls | 1 YEAR
Difference in the mean transvalvular gradient between cases and controls | 1 YEAR
Difference between maximum aortic jet velocity between cases and controls | 1 YEAR

CONTACTS AND LOCATIONS:
Locations (1):
- Fernando Civeira Murillo, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No